CLINICAL TRIAL: NCT00000377
Title: Maintenance Therapies in Late-Life Depression
Brief Title: Preventing the Return of Depression in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Charles Reynolds, Director of the Aging Institute and UPMC Endowed Professor in Geriatric Psychiatry, Neurology, and Neuroscience, University of Pittsburgh
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01MH043832 (NIH); R01MH043832 (NIH); DSIR AT-CT
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Aged; Antidepressive Agents; Depression; Dose-Response Relationship, Drug; Female; Human; Male; Middle Age; Nortriptyline; Placebos; Recurrence; Aged, 80 and over; Antidepressive Agents -- *therapeutic use; Antidepressive Agents -- administration & dosage; Depression -- *drug therapy; Nortriptyline -- *therapeutic use; Nortriptyline -- administration & dosage
MeSH Terms: conditions — Depression; Recurrence | interventions — Nortriptyline

INTERVENTIONS:
Drug: Nortriptyline

SUMMARY:
The purpose of this study is to compare the effectiveness of two doses of nortriptyline in elderly patients whose depression returned after stopping treatment. Nortriptyline is an antidepressant.

This study enrolls patients who were treated for depression in an earlier research study and whose depression has returned since stopping treatment. Patients are treated for 4 months to bring the depression under control. Patients are then assigned randomly (like tossing a coin) to receive either the full dose of nortriptyline or half the usual dose of nortriptyline. Patients continue taking nortriptyline for 2 years or until a major depression returns. Throughout the study, patients are monitored for symptoms of depression and other side effects.

DETAILED DESCRIPTION:
To determine whether elderly (60-80 years old) depressed patients who cannot sustain a remission without medication must be maintained at full acute-treatment dose. To compare the efficacy of full-dose vs half-dose nortriptyline (NT) in preventing recurrences of major depression in the elderly. To determine whether those patients who experience a recurrence while in a maintenance placebo condition (Study I) require 100 percent of their acute-treatment dose of NT to prevent subsequent recurrences or can be successfully maintained on 50 percent of their acute-treatment dose (Study II).

Investigators expect a pool of 60 patients from Study I to become eligible for Study II (the full-dose/half-dose maintenance trial). After treatment of the recurrence and following 16 weeks of stabilization therapy, patients are randomized to 1 of 2 maintenance therapy cells: full-dose NT or half-dose NT. Maintenance lasts 2 years or until recurrence of major depression. The following are assessed: differences in recurrence rates and time to recurrence under full-dose vs half-dose conditions; differences in symptomatic ratings of depression, suicidal ideation, social adjustment, and side effects; and differences in compliance rates as determined by variability in level-to-dose (L/D) ratios. Exploratory data analyses are used to generate a hypothetical profile of elderly patients who can remain well on half-dose maintenance nortriptyline.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00178100

http://clinicaltrials.gov/show/NCT00177671

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

Recurrence of major depression while in a maintenance placebo condition in the currently funded maintenance therapy protocol (Study I).

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1989-03; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Reynolds, MD, Principal Investigator

REFERENCES:
- [Result] Reynolds CF 3rd, Perel JM, Frank E, Cornes C, Miller MD, Houck PR, Mazumdar S, Stack JA, Pollock BG, Dew MA, Kupfer DJ. Three-year outcomes of maintenance nortriptyline treatment in late-life depression: a study of two fixed plasma levels. Am J Psychiatry. 1999 Aug;156(8):1177-81. doi: 10.1176/ajp.156.8.1177. PMID 10450257